CLINICAL TRIAL: NCT07266662
Title: Comparative Effects of Sensory Augmentation and Neuromodulation on Enhancing Motor Recovery Among Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/033 Asad Ali
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stroke (CVA) or Transient Ischemic Attack
Keywords: neuromuscular rehabilitation; sensory augmentation; neuromodulation; motor recovery; upper limb function; neuroplasticity; Fugl-Meyer Assessment; Jebsen-Taylor Test
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study will use a single-blind design, where the participants will be unaware of the specific intervention group they have been assigned to (i.e., whether they are receiving the combination of sensory augmentation and neuromodulation, sensory augmentation alone, or neuromodulation alone). This masking ensures that participant expectations do not influence their responses to the interventions. However, the treating therapists and study coordinators who administer the interventions and assess outcomes will not be masked, as they will be responsible for the direct management of the interventions and data collection. This design allows for an objective evaluation of the effects of the interventions while minimizing potential biases from participant expectations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (combination of Multisensory Augmentation and Neuromodulation with Routine Physical Therapy) (Experimental): Group 1 will receive a combination of Multisensory Augmentation (Mirror Therapy) and Neuromodulation (Transcranial Direct Current Stimulation - tDCS) along with Routine Physical Therapy. The interventions will be administered four times a week over an 8-week period. The multisensory augmentation component will involve Mirror Therapy, where participants will perform motor tasks with their unaffected arm while observing its reflection in a mirror placed in front of them, simulating movement of the affected arm. This therapy enhances sensory feedback and promotes neuroplasticity.
  The neuromodulation component will involve tDCS, where a low electrical current will be applied to the motor cortex to modulate cortical excitability and promote neuroplastic changes, supporting motor relearning and reducing spasticity. Each session will consist of 15 minutes of Mirror Therapy and 15 minutes of tDCS stimulation, followed by Routine Physical Therapy, which includes task-oriented training and refl
  Interventions: Other: Combination of Sensory Augmentation and Neuromodulation
- Group 2 (only sensory augmentation and Routine Physical Therapy) (Experimental): Group 2 will receive Sensory Augmentation (Mirror Therapy) in combination with Routine Physical Therapy. The interventions will be administered four times a week over an 8-week period. Mirror Therapy will involve participants performing motor tasks with their unaffected arm while observing its reflection in a mirror placed in front of them, creating the illusion of movement in the affected arm. This technique enhances sensory feedback and promotes neuroplasticity, which is critical for motor recovery in stroke survivors.
  In addition to Mirror Therapy, participants will also undergo Routine Physical Therapy for 20 minutes per session. The physical therapy will include task-oriented training and reflex inhibitory exercises designed to improve motor control, strength, and coordination. Each session will last 45 minutes, with 25 minutes dedicated to the sensory augmentation intervention and physical therapy combined. This arm aims to assess the effects of sensory augmentation alone on mot
  Interventions: Other: Sensory Augmentation
- Group 3 (neuromodulation only and Routine Physical Therapy) (Experimental): Group 3 will receive Neuromodulation (Transcranial Direct Current Stimulation - tDCS) in combination with Routine Physical Therapy. The interventions will be administered four times a week over an 8-week period. tDCS involves the application of a low electrical current to the motor cortex, modulating cortical excitability to promote neuroplasticity and support motor relearning while reducing spasticity. The tDCS session will last 20 minutes, with a 5-minute break during the session.
  In addition to tDCS, participants will also undergo Routine Physical Therapy for 20 minutes per session. The physical therapy will include task-oriented training and reflex inhibitory exercises designed to enhance motor control, strength, and functional movement. Each session will last 45 minutes, with 20 minutes dedicated to tDCS and 20 minutes to physical therapy. This arm will evaluate the impact of neuromodulation alone on motor recovery when combined with traditional physical rehabilitation techniques
  Interventions: Other: Neuromodulation

INTERVENTIONS:
Other: Sensory Augmentation — Sensory Augmentation in this study will use Mirror Therapy, a non-invasive technique aimed at enhancing sensory feedback and promoting neuroplasticity. Participants will perform tasks with their unaffected arm while observing its reflection in a mirror placed in front of them, creating the illusion that the affected arm is moving. This visual feedback stimulates sensory pathways and encourages the brain to reorganize motor functions. Each session will last 15 minutes, conducted four times a week for 8 weeks, alongside Routine Physical Therapy. Mirror therapy differs from other rehabilitation methods by focusing on sensory-motor deficits through visual feedback, encouraging neuroplasticity and motor recovery, especially in chronic stroke patients with upper limb impairments.
  Other Names: Routine Physical Therapy
  Arms: Group 2 (only sensory augmentation and Routine Physical Therapy)
Other: Neuromodulation — Neuromodulation in this study will use Transcranial Direct Current Stimulation (tDCS), a non-invasive technique to modulate brain activity. A low electrical current will be applied to the motor cortex to enhance cortical excitability, promote neuroplasticity, and support motor relearning. tDCS helps reduce spasticity and facilitates recovery of motor functions by altering neural activity in targeted areas of the brain. Each session will last 20 minutes, with a 5-minute break, conducted four times a week for 8 weeks, alongside Routine Physical Therapy. tDCS stands apart from other therapies by directly stimulating brain regions to enhance neural plasticity, targeting motor function recovery through brain stimulation rather than external physical exercises alone.
  Other Names: Routine Physical Therapy
  Arms: Group 3 (neuromodulation only and Routine Physical Therapy)
Other: Combination of Sensory Augmentation and Neuromodulation — The combined intervention will integrate Transcranial Direct Current Stimulation (tDCS) and Mirror Therapy to enhance motor recovery through both brain stimulation and sensory feedback. tDCS will apply a low electrical current to the motor cortex to modulate brain activity, promoting neuroplasticity, reducing spasticity, and facilitating motor relearning. Mirror Therapy will provide visual feedback by having participants perform tasks with their unaffected arm while observing its reflection in a mirror, simulating movement in the affected arm and stimulating sensory-motor pathways. This combined approach aims to maximize neuroplasticity by targeting both the brain and sensory processing systems. Each session will last 45 minutes: 15 minutes of Mirror Therapy, 15 minutes of tDCS, and 15 minutes of Routine Physical Therapy, conducted four times a week for 8 weeks.
  Other Names: Routine Physical Therapy
  Arms: Group 1 (combination of Multisensory Augmentation and Neuromodulation with Routine Physical Therapy)

SUMMARY:
This study aims to evaluate the effectiveness of two rehabilitation techniques-Sensory Augmentation (using mirror therapy) and Neuromodulation (using transcranial direct current stimulation, tDCS)-in improving motor recovery among stroke survivors. Stroke often results in long-term impairments, particularly in upper limb motor function, which is critical for daily activities. Although current rehabilitation strategies help, more effective solutions are needed to enhance recovery. Participants, aged 45-65 with chronic stroke and upper extremity impairments, will be randomized into three groups: Group 1 will receive a combination of sensory augmentation (mirror therapy) and neuromodulation (tDCS) with routine physical therapy; Group 2 will receive sensory augmentation (mirror therapy) with routine physical therapy; and Group 3 will receive neuromodulation (tDCS) with routine physical therapy. The interventions will take place four times a week for 8 weeks, and participants will undergo motor function assessments, including the Fugl-Meyer Assessment and Jebsen-Taylor Test, before and after the intervention. The study will compare the effects of each intervention on motor recovery, specifically focusing on upper limb function and motor control. The findings could lead to improved rehabilitation protocols, offering stroke survivors better therapeutic options and enhancing their quality of life.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of disability worldwide, often leading to long-term impairments in motor function, particularly in the upper limbs. These impairments can severely affect a person's ability to perform daily tasks, reducing their independence and quality of life. The rehabilitation process for stroke survivors typically includes physical therapy aimed at improving motor control, balance, and functionality of the affected limbs. While traditional rehabilitation strategies are effective, there is a growing interest in enhancing recovery through advanced techniques such as Sensory Augmentation and Neuromodulation.

This study will focus on evaluating the comparative effects of two innovative rehabilitation approaches-Sensory Augmentation through Mirror Therapy and Neuromodulation through Transcranial Direct Current Stimulation (tDCS)-on motor recovery in chronic stroke survivors. These two techniques have shown promising results in improving motor function in stroke patients, but their combined effect remains unclear.

Intervention Strategies:

Sensory Augmentation: Mirror therapy is a non-invasive technique that involves using a mirror to create the illusion of movement in the affected limb by reflecting the movement of the unaffected limb. This process enhances the sensory feedback and promotes neuroplasticity, which is the brain's ability to reorganize and form new neural connections. Mirror therapy has been shown to reduce spasticity, improve sensory functions like proprioception, and facilitate the restoration of motor function.

Neuromodulation: Transcranial Direct Current Stimulation (tDCS) is a non-invasive brain stimulation technique that uses a low electrical current to modulate neuronal activity in specific areas of the brain. For stroke survivors, tDCS is applied to the motor cortex to promote neuroplasticity, facilitate the relearning of motor tasks, and reduce spasticity. While previous studies have demonstrated the effectiveness of tDCS, its impact when combined with sensory augmentation has not been fully explored.

Study Design and Groups:

This randomized controlled trial will involve 36 chronic stroke patients aged 45-65 who have upper extremity motor impairments. The participants will be randomly assigned to one of three groups:

Group 1 (Experimental Group): A combination of sensory augmentation (mirror therapy) and neuromodulation (tDCS) along with routine physical therapy.

Group 2: Sensory augmentation (mirror therapy) combined with routine physical therapy.

Group 3: Neuromodulation (tDCS) combined with routine physical therapy.

Each participant will undergo the interventions four times a week for 8 weeks. Routine physical therapy will include task-oriented training and reflex inhibitory patterns exercises aimed at improving motor control and coordination. Both sensory augmentation and neuromodulation will be administered for 30 minutes per session, with each intervention lasting 15 minutes for mirror therapy and 15 minutes for tDCS. The entire session, including physical therapy, will last for 45 minutes.

Outcome Measures:

The primary outcome of the study will be the improvement in upper limb motor function, measured by the Fugl-Meyer Assessment (FMA) for motor function and the Jebsen-Taylor Test, which assesses functional hand tasks. These assessments will be conducted before the intervention, at 4 weeks, and at 8 weeks to evaluate both short-term and long-term effects.

Secondary outcomes will include improvements in the quality of life, as measured by validated scales like the Stroke Impact Scale (SIS), and the impact on daily activities, such as handgrip strength, motor coordination, and task performance. The effects on spasticity and sensory function will also be monitored.

Data Collection and Analysis:

Data will be collected at multiple time points during the study to assess the effects of the interventions on motor function, spasticity, and quality of life. Statistical analyses will include mixed-model ANOVA to examine the effects of time and intervention group on the primary and secondary outcomes. Post-intervention comparisons will be made to assess the differential impact of each intervention. Additionally, repeated measures ANOVA will be conducted to track within-group improvements over time.

Safety and Ethics:

This study has been approved by the institutional review board (IRB) of Lahore University of Biological and Applied Sciences, and all participants will provide informed consent before participating. To ensure the safety of participants, all sessions will be conducted under the supervision of trained physical therapists. Minimal risks associated with the study include mild discomfort or fatigue during the physical assessments and interventions. If any participant experiences adverse effects, they will be promptly withdrawn from the study.

The study will also ensure the confidentiality of all participant data. Personal information will be anonymized, and data will be stored securely. Participation in the study is voluntary, and participants may withdraw at any time without facing any negative consequences.

Significance and Potential Impact:

This study has the potential to significantly impact stroke rehabilitation practices by providing evidence on the comparative efficacy of sensory augmentation and neuromodulation techniques in enhancing motor recovery. The results may guide clinicians in developing more effective rehabilitation protocols and inform future research on combined rehabilitation strategies.

Given the growing incidence of stroke worldwide, particularly in low- and middle-income countries, this research could pave the way for accessible, cost-effective, and non-invasive therapeutic interventions. It may offer stroke survivors, especially those in resource-limited settings, improved chances for motor recovery and a better quality of life. Furthermore, this study will contribute valuable data to the scientific community, offering insights into the combined effects of mirror therapy and tDCS, which could enhance the evidence base for stroke rehabilitation.

Conclusion:

By comparing the effects of sensory augmentation and neuromodulation, this study aims to identify the most effective intervention(s) for improving motor recovery in stroke survivors. The findings will not only contribute to the field of neurorehabilitation but may also offer new therapeutic options for patients in need of effective, evidence-based treatments for motor impairments post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-65
* Gender: both male and female
* Ischemic stroke
* Diagnosed cases of middle cerebral artery stroke by neurologist
* Stage of recovery - Chronic (more than 6 months)
* Burnstromm recovery stage 3
* Good Compliance

Exclusion Criteria:

* Vestibular Dysfunction
* Serious cognitive impairment,
* Severe vision or visuospatial neglect
* Spasticity (Modified Ashworth scale >3)
* Upper extremity contractures
* Upper extremity fractures
* Orthopedic disease
* Neurological conditions (other than stroke)
* Recurrence of stroke or epilepsy during the study period
* Serious systemic impairment or concomitant diseases
* Patients refused to participate in the experiment

Ages: 45 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale | Primary and secondary outcome measures will be assessed at baseline, 4 weeks, and 8 weeks to track changes in motor recovery and functional abilities.
  The Fugl-Meyer Assessment (FMA) is a comprehensive, standardized tool used to assess motor function recovery in stroke patients, focusing on the upper limb, balance, and sensory function. The FMA includes subscales for motor function, sensory function, balance, and joint range of motion. The motor function subscale, which is particularly relevant in this study, evaluates voluntary movements, reflexes, coordination, and muscle strength of the upper limbs.
  The FMA scale ranges from 0 to 66 for the upper limb, with higher scores indicating better motor function. A score of 66 represents full motor recovery, while 0 indicates no motor function. Intermediate scores reflect varying levels of impairment and recovery. The FMA is widely used for its sensitivity in detecting changes over time, making it an effective tool for tracking motor recovery after stroke.
Jebsen-Taylor Test | Primary and secondary outcome measures will be assessed at baseline, 4 weeks, and 8 weeks to track changes in motor recovery and functional abilities.
  The Jebsen-Taylor Test of Hand Function (JTT) is a standardized assessment used to evaluate the functional use of the hands in everyday tasks, particularly for stroke patients. It includes seven subtests: writing, card turning, picking up small objects, simulated feeding, stacking checkers, and moving light and heavy objects. These tasks simulate common daily activities that require hand function.
  The JTT is scored based on the time it takes to complete each task, with shorter times indicating better hand function. The total score is the sum of the times for all subtests. Interpretation: Lower total times suggest better hand function, while longer times indicate greater motor impairment. The test helps assess the ability to perform functional tasks, providing a realistic measure of hand performance and recovery. It's valuable for evaluating improvements in motor function following rehabilitation interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Nabeela Dawood, Study Chair — Lahore University of Biological and Applied Sciences
Locations (2):
- Pakistan (2):
  - Lahore University of Biological and Applied Sciences, Lahore, Punjab Province
  - Pakistan Society of Rehabilitation and Differently Abled Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahid J, Kashif A, Shahid MK. A Comprehensive Review of Physical Therapy Interventions for Stroke Rehabilitation: Impairment-Based Approaches and Functional Goals. Brain Sci. 2023 Apr 25;13(5):717. doi: 10.3390/brainsci13050717. PMID 37239189
- [Background] Norman SL, Wolpaw JR, Reinkensmeyer DJ. Targeting neuroplasticity to improve motor recovery after stroke: an artificial neural network model. Brain Commun. 2022 Oct 21;4(6):fcac264. doi: 10.1093/braincomms/fcac264. eCollection 2022. PMID 36458210
- [Background] Harris JE, Eng JJ. Paretic upper-limb strength best explains arm activity in people with stroke. Phys Ther. 2007 Jan;87(1):88-97. doi: 10.2522/ptj.20060065. Epub 2006 Dec 19. PMID 17179441
- [Background] Li S. Spasticity, Motor Recovery, and Neural Plasticity after Stroke. Front Neurol. 2017 Apr 3;8:120. doi: 10.3389/fneur.2017.00120. eCollection 2017. PMID 28421032
- [Background] Coupland AP, Thapar A, Qureshi MI, Jenkins H, Davies AH. The definition of stroke. J R Soc Med. 2017 Jan;110(1):9-12. doi: 10.1177/0141076816680121. Epub 2017 Jan 13. No abstract available. PMID 28084167